CLINICAL TRIAL: NCT05012605
Title: The SLEEPR Study: SLEep Effects on Post-stroke Rehabilitation
Acronym: SLEEPR
Status: Recruiting | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Karen J. Klingman PhD RN, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: R01NR018979 (NIH)
Record Dates: First submitted 2021-08-09; First posted 2021-08-19 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Sleep Wake Disorders; Rehabilitation; Recovery of Function
Keywords: Longitudinal study; actigraphy; spatial analysis; patient reported outcome measures; wearable electronic devices
MeSH Terms: conditions — Stroke; Sleep Wake Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLEEPR cohort: Individuals within first 3 months following stroke who did not have obstructive sleep apnea within the first 15 days following stroke
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observe physical function and sleep disorder symptoms following stroke

SUMMARY:
Sleep is critical for health and quality of life; however, little is known about the prevalence or impact of non obstructive sleep apnea (non-OSA) sleep disorders in people with stroke. The proposed study aims to characterize the proportion of people with stroke that have non-OSA sleep disorders and their impact on recovery of activities of daily living, functional mobility, and participation along the continuum of recovery in people with stroke.

DETAILED DESCRIPTION:
The overall goal in this project is to develop an in-depth understanding of the complex interplay between non-obstructive sleep apnea (non OSA) sleep disorders and recovery after stroke. Sleep is vital to overall health and quality of life. Abnormal or insufficient sleep is both a risk factor and consequence of stroke. Sleep also plays a critical role in motor learning, which is the foundation of rehabilitation strategies after stroke. Although there is a growing understanding of the interplay between sleep, stroke, and recovery in people with OSA these complex relationships in individuals post stroke with non OSA sleep disorders are not well understood. In order to develop targeted sleep interventions to support rehabilitation after stroke and promote optimal recovery, it is critical to gain a fuller understanding of the prevalence and impact of non OSA sleep disorders in people with stroke across the continuum of recovery. The specific objectives of this proposal will lay the necessary groundwork for this as investigators will characterize the proportion of people with stroke that have insomnia disorders, restless legs syndrome, and insufficient sleep; and evaluate the impact of these non OSA sleep disorders on recovery of activities of daily living, mobility/activity, and participation across the continuum of recovery after stroke. The study will take an innovative approach to measuring sleep, mobility/activity, and participation using a combination of techniques across the measurement spectrum that will include self-report questionnaires, clinic-based measures of capacity, and body worn sensors. The body worn sensors will include actigraphy to measure sleep parameters, activity monitors to measure mobility/activity levels, and Global Positioning System (GPS) units to measure participation. Additionally, investigators will apply innovative, big data tools from topological data analysis for a data driven approach to discover complex, structural, non-linear interdependent relationships among stroke, sleep, and recovery of mobility/activity, and participation. Upon completion of this study there will be an understanding of the prevalence and impact of non-OSA sleep disorders on recovery of function, mobility/activity, and participation across the continuum of recovery post stroke. This is an important, necessary step to develop appropriate sleep-based interventions to complement targeted rehabilitation strategies to enhance the health and quality of life in people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke as defined by the WHO: "a rapid onset event of vascular origin reflecting a focal disturbance of cerebral function, excluding isolated impairments of higher function and persisting longer than 24 hours." Diagnosis of stroke will be confirmed by imaging or clinical diagnosis.
* Age 18 or older.
* Admitted to in-patient rehabilitation.
* National Institutes of Health Stroke Scale (NIHSS) item 1a score <2 (Level of consciousness: 0=alert, 1=not alert, but arousable by minor stimulation to obey, answer, or respond).
* Provision of informed consent by individual or by legally authorized representative.

Exclusion Criteria:

* Pre-stroke or current diagnosis of OSA or other sleep-related breathing disorder.
* Living in a nursing home or assisted living center prior to the stroke.
* Unable to ambulate 150' independently prior to the stroke.
* Other neurologic health condition that may impact recovery such as Parkinson Disease, Multiple Sclerosis, Traumatic Brain Injury, Alzheimer's Disease.
* Women who are pregnant.
* Recent hemicraniectomy or suboccipital craniectomy (i.e. those whose bone has not yet been replaced), or any other recent bone removal procedure for relief of intracranial pressure.
* Planned discharge location >150 miles radius from recruitment site
* Global aphasia as defined by a NIHSS item 9 score of 3 (3= Mute, global aphasia; no usable speech or auditory comprehension).
* Inability to understand English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults recovering from stroke within the first 90 days following stroke who did not have a diagnosis of obstructive sleep apnea (OSA) prior to stroke or who do not have oxygen desaturation index (ODI) of 15 or higher during inpatient rehabilitation (~15 days post-stroke).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional independence with activities of daily living as measured by the Barthel index | 15 days post-stroke
  The Barthel index is a measure of functional independence with activities of daily living; the score range is 0-100 with higher numbers indicating more independence
Functional independence with activities of daily living as measured by the Barthel index | 60 days post-stroke
  The Barthel index is a measure of functional independence with activities of daily living; the score range is 0-100 with higher numbers indicating more independence
Functional independence with activities of daily living as measured by the Barthel index | 90 days post-stroke
  The Barthel index is a measure of functional independence with activities of daily living; the score ranges 0-100 with higher numbers indicating more independence
Level of disability according to the stroke impact scale | 60 days post-stroke
  The stroke impact scale is a self-report measure of disability; scores range from 0-100 with higher numbers indicating better function
Level of disability according to the stroke impact scale | 90 days post-stroke
  The stroke impact scale is a self-report measure of disability; scores range from 0-100 with higher numbers indicating better function
Daytime sleepiness according to the Epworth Sleepiness Scale | 15 days post-stroke
  Epworth sleepiness scale is a self report measure describing likelihood of falling asleep during different circumstances; scores range from 0-24, with higher numbers indicating more sleepiness
Daytime sleepiness according to the Epworth Sleepiness Scale | 60 days post-stroke
  Epworth sleepiness scale is a self report measure describing likelihood of falling asleep during different circumstances; scores range from 0-24, with higher numbers indicating more sleepiness
Daytime sleepiness according to the Epworth Sleepiness Scale | 90 days post-stroke
  Epworth sleepiness scale is a self report measure describing likelihood of falling asleep during different circumstances; scores range from 0-24, with higher numbers indicating more sleepiness
Insomnia severity as determined from the insomnia severity index | 15 days post-stroke
  The insomnia severity index is a self report measure of insomnia severity; scores range from 0-28, with higher numbers indicating more severe insomnia
Insomnia severity as determined from the insomnia severity index | 60 days post-stroke
  The insomnia severity index is a self report measure of insomnia severity; scores range from 0-28, with higher numbers indicating more severe insomnia
Insomnia severity as determined from the insomnia severity index | 90 days post-stroke
  The insomnia severity index is a self report measure of insomnia severity; scores range from 0-28, with higher numbers indicating more severe insomnia
Likely presence of restless legs syndrome as measured by the Cambridge Hopkins restless legs questionnaire | 15 days post-stroke
  The Cambridge Hopkins restless legs questionnaire is a self report measure of presence and frequency of symptoms of restless legs syndrome; responses are scored according to an algorithm that provides yes/no for likely presence of restless legs syndrome.
Likely presence of restless legs syndrome as measured by the Cambridge Hopkins restless legs questionnaire | 60 days post-stroke
  The Cambridge Hopkins restless legs questionnaire is a self report measure of presence and frequency of symptoms of restless legs syndrome; responses are scored according to an algorithm that provides yes/no for likely presence of restless legs syndrome.
Likely presence of restless legs syndrome as measured by the Cambridge Hopkins restless legs questionnaire | 90 days post-stroke
  The Cambridge Hopkins restless legs questionnaire is a self report measure of presence and frequency of symptoms of restless legs syndrome; responses are scored according to an algorithm that provides yes/no for likely presence of restless legs syndrome.
Cumulative morbidity of sleep disorders, as determined from the sleep disorders checklist, 25 item version | 15days post-stroke
  The sleep disorders checklist, 25 item version, is a self report questionnaire of frequency of occurrence of 25 sleep disorder symptoms; scores range from 0-100, with higher numbers indicating worse overall morbidity of sleep disorders.
Cumulative morbidity of sleep disorders, as determined from the sleep disorders checklist, 25 item version | 60days post-stroke
  The sleep disorders checklist, 25 item version, is a self report questionnaire of frequency of occurrence of 25 sleep disorder symptoms; scores range from 0-100, with higher numbers indicating worse overall morbidity of sleep disorders.
Cumulative morbidity of sleep disorders, as determined from the sleep disorders checklist, 25 item version | 90 days post-stroke
  The sleep disorders checklist, 25 item version, is a self report questionnaire of frequency of occurrence of 25 sleep disorder symptoms; scores range from 0-100, with higher numbers indicating worse overall morbidity of sleep disorders.

SECONDARY OUTCOMES:
Degree of disability according to the modified Rankin scale | 15 days post-stroke
  the modified Rankin scale is used to measure degree of disability in patients who have had a stroke; scores range from 0-5, with higher numbers indicating the most disability
Degree of disability according to the modified Rankin scale | 60 days post-stroke
  the modified Rankin scale is used to measure degree of disability in patients who have had a stroke; scores range from 0-5, with higher numbers indicating the most disability
Degree of disability according to the modified Rankin scale | 90 days post-stroke
  the modified Rankin scale is used to measure degree of disability in patients who have had a stroke; scores range from 0-5, with higher numbers indicating the most disability
Balance ability according to the Berg balance scale | 15 days post-stroke
  The Berg balance scale is an observational measure of balance ability according to performance on 14 tasks; scores range from 0-56, with higher scores indicating better balance
Balance ability according to the Berg balance scale | 60 days post-stroke
  The Berg balance scale is an observational measure of balance ability according to performance on 14 tasks; scores range from 0-56, with higher scores indicating better balance
Balance ability according to the Berg balance scale | 90 days post-stroke
  The Berg balance scale is an observational measure of balance ability according to performance on 14 tasks; scores range from 0-56, with higher scores indicating better balance
Gait speed | 15 days post-stroke
  Objective measure of gait speed from 10 meter walk test
Gait speed | 60 days post-stroke
  Objective measure of gait speed from 10 meter walk test
Gait speed | 90 days post-stroke
  Objective measure of gait speed from 10 meter walk test
Activity level | 15 days post-stroke
  Objective measure of activity according to leg-worn activity monitor to be analyzed according to manufacturer's algorithm.
Activity level | 60 days post-stroke
  Objective measure of activity according to leg-worn activity monitor to be analyzed according to manufacturer's algorithm.
Activity level | 90 days post-stroke
  Objective measure of activity according to leg-worn activity monitor to be analyzed according to manufacturer's algorithm.
Types of community locations visited by study participants, as determined from global positioning sensor data | 60 days post-stroke
  Objective measure of location of participant over a one week timeframe
Types of community locations visited by study participants, as determined from global positioning sensor data | 90 days post-stroke
  Objective measure of location of participant over a one week timeframe
GG code for Mobility and Self Care Sections | 15 days post-stroke
  Self care and functional mobility codes extracted from participants' medical records
Daily activities as recorded by study participants (trip log) | 60-days post-stroke
  tabulation of trip log - record of when they leave the house and where they are going.
Daily activities as recorded by study participants (trip log) | 90-days post-stroke
  tabulation of trip log - record of when they leave the house and where they are going.
Cognitive ability according to the Montreal cognitive assessment | 15 days post-stroke
  the Montreal cognitive assessment ratess participants' performance on several tasks as scored by a trained observer; scores range 0-30 with higher scores indicating better cognitive ability.
Cognitive ability according to the Montreal cognitive assessment | 60 days post-stroke
  the Montreal cognitive assessment ratess participants' performance on several tasks as scored by a trained observer; scores range 0-30 with higher scores indicating better cognitive ability.
Cognitive ability according to the Montreal cognitive assessment | 90 days post-stroke
  the Montreal cognitive assessment ratess participants' performance on several tasks as scored by a trained observer; scores range 0-30 with higher scores indicating better cognitive ability.
Depression severity as measured by the patient health questionnaire (9-item version) | 15 days post-stroke
  This is a self-report scale measuring frequency of depressive symptoms; scores range from 0-27 with higher scores indicating more severe depression
Depression severity as measured by the patient health questionnaire (9-item version) | 60 days post-stroke
  This is a self-report scale measuring frequency of depressive symptoms; scores range from 0-27 with higher scores indicating more severe depression
Depression severity as measured by the patient health questionnaire (9-item version) | 90 days post-stroke
  This is a self-report scale measuring frequency of depressive symptoms; scores range from 0-27 with higher scores indicating more severe depression
Sleep diary | 60 days post-stroke
  Tabulation of participant's sleep habits from a written diary, over a one week timeframe.
Sleep diary | 90 days post-stroke
  Tabulation of participant's sleep habits from a written diary, over a one week timeframe.
Oxygen desaturation index | 90 days post-stroke
  Oxygen desaturations per minute index, as determined from a pulse oximeter worn overnight
Oxygen desaturation index | 60 days post-stroke
  Oxygen desaturations per minute index, as determined from a pulse oximeter worn overnight
Oxygen desaturation index | 15 days post-stroke
  Oxygen desaturations per minute index, as determined from a pulse oximeter worn overnight
Wrist actigraphy data | 15 days post-stroke
  Data measured from a wrist-worn actigraph, to be analyzed according to manufacturer's algorithm
Wrist actigraphy data | 60 days post-stroke
  Data measured from a wrist-worn actigraph, to be analyzed according to manufacturer's algorithm
Wrist actigraphy data | 90 days post-stroke
  Data measured from a wrist-worn actigraph, to be analyzed according to manufacturer's algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Klingman, PhD, Principal Investigator — SUNY Upstate Medical University, College of Nursing
Locations (6):
- United States (6):
  - Emory University, Atlanta, Georgia
  - KU Medical Center, The University of Kansas, Kansas City, Kansas
  - Institute for Human Performance - Upstate Rehabilitation at IHP, Syracuse, New York
  - Upstate University Hospital, Syracuse, New York
  - Upstate Community Hospital, Syracuse, New York
  - Good Shepherd Rehabilitation Network, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Final research data along with meta-data and descriptors will be shared to the maximum extent possible while protecting patient privacy. Data will be for individual subjects. No aggregate data will be provided apart from what is published in the literature. Data will be formatted for SPSS and/or as csv files.
Supporting Information: Study Protocol
Time Frame: Anticipated availability of the dataset will be announced during the final year of the project, with notification of how to apply for access to the data. Data will be deposited into the institutional repository as soon as possible, after key manuscripts have been accepted for publication. Should manuscripts be delayed due to unforeseen circumstances, data will be available through the repository within a year of project closure. Data will remain available by request from the PI during time of employment at SUNY Upstate, after which time the SUNY Upstate library will manage and grant access according to guidelines set forth by the IRB.
Access Criteria: An online data request form will be available so that others can indicate their interest in the data through a publicly available website. A data sharing agreement will be signed by all parties.
  Because detailed pattern of life information may contain information that may allow subject identity to be recovered, we intend to provide two levels of data sharing with three classes of data.
  1. Controlled share: data (to include pattern-of-life data) that contains information for which identity could be recovered if analyzed with malicious intent. These data will only be released to vetted researchers under conditions that provide assurance of protected privacy.
  2. Public share: a subset of the variables that are not expected to provide privacy risk; and Geo-summarized or modified data - consistent with state-of-the-art methodologies for differential privacy, the collected participation (geolocation) data will be made available after the data has been modified to preserve privacy.

REFERENCES:
- [Derived] Klingman KJ, Skufca JD, Duncan PW, Wang D, Fulk GD. Study Protocol: Sleep Effects on Poststroke Rehabilitation Study. Nurs Res. 2022 Nov-Dec 01;71(6):483-490. doi: 10.1097/NNR.0000000000000611. Epub 2022 Aug 6. PMID 35948301